CLINICAL TRIAL: NCT00994552
Title: A Pilot Study: Comparing Physiological Parameters and Outcome Variables Using Pressure Support Ventilation Versus Pressure Controlled Ventilation in Patients With Chronic Respiratory Failure
Brief Title: Comparison of Pressure Support and Pressure Control Ventilation in Chronic Respiratory Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Karen Ignathian, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 09/H0802/3
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: COPD; Chest Wall Disease; Neuromuscular Disease; Obesity Hypoventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure support ventilation (Active Comparator): Pressure support ventilation
  Interventions: Other: Pressure support ventilation
- Pressure control ventilation (Active Comparator): Pressure control ventilation
  Interventions: Other: Pressure control ventilation

INTERVENTIONS:
Other: Pressure support ventilation — Pressure support ventilation
  Arms: Pressure support ventilation
Other: Pressure control ventilation — Pressure control ventilation
  Arms: Pressure control ventilation

SUMMARY:
This study is looking at whether there is a difference in outcomes using two different types of breathing support in those patients who have chronic respiratory failure (patients who under-breathe).

There is little data to demonstrate which mode of ventilation is better in terms of physiological outcomes and outcome data relating to patient symptoms.

We hypothesize that one type of breathing support: pressure support ventilation would be more comfortable for patients as it more closely matches a patient's own respiratory pattern and and so leads to improved adherence and consequent improvement in quality of life.

Patients with respiratory failure will be randomly assigned to receive either pressure support ventilation or pressure control ventilation for the first 6 weeks and then cross-over to receive the mode not previously used for a further 6 weeks. They will have baseline data recorded and then be followed up after each 6 week block.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest wall deformity, neuromuscular disease or obesity hypoventilation syndrome with an FEV1/FVC ratio of >70% and VC <50% predicted or patients with COPD with a FEV1/FVC ratio of <70% an FEV1 <50% predicted
* Stable

  * pH >7.35
  * ESS <18
  * Symptomatically stable with clinical resolution of intercurrent infection: normal C reactive protein, white cell count and afebrile
* Daytime symptoms compatible with nocturnal hypoventilation i.e. poor sleep, morning headache, daytime somnolence, shortness of breath
* Arterial carbon dioxide partial pressure (PaCO2) > 6.0kPa during day with evidence of nocturnal hypoventilation (TcCO2 >7.5KPa or a rise in TcCO2 of >1 KPa)
* No prior domiciliary ventilation use
* Patients with COPD must be established on optimal medical treatment prior to enrolment

Exclusion Criteria:

* Psychological, social or geographical situation that would impair compliance with the schedule
* Patients who have underlying malignancy or severe cardiac dysfunction (ejection fraction <40%)
* Complex OSA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Adherence to ventilation | 6 and 12 weeks

SECONDARY OUTCOMES:
Arterial blood gases | 6 and 12 weeks
Health related quality of life as measured by CRQ and SRI | 6 and 12 weeks
Breathlessness (MRC dyspnoea score) | 6 and 12 weeks
Assessment of daytime vigilance and fatigue by the Epworth sleepiness score,Oxford sleep resistance test and the fatigue severity score. | 6 and 12 weeks
Sleep comfort as assessed by a visual analogue scale | 6 and 12 weeks
Spirometry: forced expiratory volume in 1s and forced vital capacity | 6 and 12 weeks
Respiratory muscle strength: maximum inspiratory pressure, maximum expiratory pressure and sniff nasal pressure | 6 and 12 weeks
Sleep fragmentation as assessed by actigraphy | 2 week perids from 4 and 10 weeks
Patient ventilator synchrony as measured by number of ineffective efforts | 6 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A Davidson, MA, MD, Study Chair — Guys's and St Thomas' NHS foundation trust; N Hart, MB BS, PhD, Principal Investigator — Guy's and St Thomas' Foundation Trust; K Brignall, MB ChB, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Murphy PB, Brignall K, Moxham J, Polkey MI, Davidson AC, Hart N. High pressure versus high intensity noninvasive ventilation in stable hypercapnic chronic obstructive pulmonary disease: a randomized crossover trial. Int J Chron Obstruct Pulmon Dis. 2012;7:811-8. doi: 10.2147/COPD.S36151. Epub 2012 Dec 11. PMID 23271905